CLINICAL TRIAL: NCT05151900
Title: Understanding and Mitigating the Impact of the COVID-19 Pandemic on Children, Youth, and Families Living With an Eating Disorder: A National Implementation Study of a Virtual Parent-Led Peer Support Intervention
Brief Title: Implementing Virtual Parent Support Groups for Eating Disorders Across Canada
Acronym: vPLPSG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jennifer Couturier, Principal Investigator, Medical Co-Director, Associate Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14196
Record Dates: First submitted 2021-10-29; First posted 2021-12-09 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Eating Disorders
Keywords: eating disorder; parent support group; COVID-19
MeSH Terms: conditions — Feeding and Eating Disorders; COVID-19 | interventions — Self-Help Groups; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stakeholder Perspectives and Virtual Parent-Led Peer Support Group (Experimental): Qualitative interviews regarding the impact of COVID-19 will be conducted with youth who have an eating disorder (ED), parents of youth who have an ED, ED clinicians and ED program administrators, as well as get their perspectives on parent-led peer support groups. Three parent-led peer support groups will be started, including psychoeducation in a virtual group setting for parents who have a child or adolescent with an eating disorder.
  Interventions: Behavioral: Support Group for Caregivers

INTERVENTIONS:
Behavioral: Support Group for Caregivers — Engage parents in the community via this support group, so they can be supported by other parents who "know the system", can advise them on how to proceed, and empower them to help their children. Parents will learn psychoeducation about eating disorders and how to support their children.

SUMMARY:
During the COVID-19 pandemic, Canada has experienced a surge in new pediatric eating disorder cases and hospitalizations and long treatment waitlists, with parents experiencing anxiety due to a lack of support. As it has not been rigorously studied, there is an urgent need to understand and mitigate the impact of the COVID-19 pandemic on children, youth, and families living with eating disorders across Canada. The investigator's proposed research has two goals. First, the investigators plan to understand the impact of the COVID-19 pandemic faced by this population throughout the country, as well as describe stakeholder views on virtual parent-led peer support groups. Given the increased burden faced by parents of children with eating disorders during the COVID-19 pandemic, the second goal is to study whether the national implementation of virtual parent-led peer support groups helps to mitigate the impact of the pandemic among affected parents. The investigators will use qualitative semi-structured interviews to gather an understanding of the impact of the pandemic on relevant stakeholders across the country. At the same time, the investigators will evaluate the feasibility and acceptability of the implementation of virtual parent-led peer support groups in several regions of Canada by examining parent and parent peer support provider experiences.

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to write, speak and understand English
* Have access to a computer and internet
* Among parents enrolled in the virtual parent-led peer support groups, they must have a child or adolescent (<18 years of age) diagnosed with an eating disorder
* Among youth and parents of youth with an eating disorder in the qualitative interviews component of the study, they/their child must either be on a waiting list for eating disorder treatment, actively in treatment, or post-treatment; the youth must be <18 years of age and the parent must have a child <18 years of age
* Among clinician/administrators in the qualitative interviews component of the study, they must work within pediatric eating disorder programs or lifespan eating disorder programs.

Exclusion Criteria:

* No lived or professional experience in the field of eating disorders
* Don't have the capacity to write, speak and understand English
* Don't have access to the internet/computer

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Parent, youth, clinician, and administrator perspectives on and experiences with the COVID-19 pandemic and children, youth, and families with eating disorders | Baseline to 6 months later
  Perspectives and experiences qualitatively measured by semi-structured individual interviews with participants with lived experience or expertise in pediatric eating disorders during the COVID-19 pandemic.
Parent, youth, clinician, and administrator perspectives on virtual parent-led peer support groups to help mitigate the negative effects of COVID-19 on children, youth, and families with eating disorders across Canada | Baseline to 6 months later
  Perspectives qualitatively measured by semi-structured individual interviews with participants with lived experience or expertise in pediatric eating disorders during the COVID-19 pandemic.
Parent, youth, clinician, and administrator perspectives on factors important for implementing and sustaining virtual parent-led peer support groups | Baseline to 6 months later
  Perspectives qualitatively measured by semi-structured individual interviews with participants with lived experience or expertise in pediatric eating disorders during the COVID-19 pandemic.

SECONDARY OUTCOMES:
Change in number of parents who remain in the support group (Retention Rate) | Baseline and 3 months later
  The investigators will compare the number of parents who consent to participate in the support group and study to the number of parents who have completed the support group and study, 3 months later.
Number of support groups each parent attends (Attendance Rate) | 3 months after baseline
  The investigators will take note of how many support groups (out of 6) each parent attends in a 3 month period.
Change in self-reported parental burden | Baseline and 3 months later
  Parental burden will be assessed using the Eating Disorders Symptom Impact Scale (EDSIS) - a 24 item measure examining the impact of symptoms on parents' lives. Minimum score is 0, maximum score is 96. A higher score indicates that the child's eating disorder symptoms are having a greater impact on their parent (more burdensome).
Change in self-reported needs as a parent of a child with an eating disorder | Baseline and 3 months later
  Parental needs will be assessed using the Carers Needs Assessment Measure (CaNAM), a 47-item questionnaire examining information received about eating disorders, support received from other people and organizations, support for self, and areas where help is needed. The minimum score is 0, the maximum score is 64. A higher score indicates that the carer has received sufficient information and support for themselves and their child.
Change in self-reported parental self efficacy and collaboration | Baseline and 3 months later
  Parental self-efficacy and collaboration will be assessed using the Patient and Carer Collaboration Scale -C (PACCS), a 33-item questionnaire examining constructs such as hope, self-care and compassion, externalization of the eating disorder, and boundaries. Each question is evaluated on a scale of 0 to 100, where higher values indicate positive collaboration with their child and higher parental self efficacy.
Parent Peer Support Providers' Change in Readiness | Baseline and 6 months later
  The Brief Individual Readiness to Change Scale will indicate how ready parent peer support providers feel they are to change. Higher scores indicate greater readiness to use research-based direct service techniques. Minimum score is 0, maximum score is 20.
Parent Peer Support Providers' Change in Attitudes about Evidence Based Practice | Baseline and 6 months later
  Their attitudes about evidence-based practice will be assessed using the Evidence Based Practice Attitudes Scale (EBPAS). The subscales include requirements, appeal, openness and divergence. The score for each subscale is created by computing a mean score for the items that load on a given subscale. Minimum score for each subscale is 0, maximum score for each subscale is 4.
Parent Peer Support Providers' Change in Confidence related to the Intervention | Baseline and 6 months later
  Their confidence related to the intervention will be assessed by administering an adapted version of the Perceived Attributes of the Principles of Effectiveness Scale (MPAS). Higher scores are indicative of more favorable perception for virtual parent led peer support group content. The minimum score is 18, the maximum score is 90.
Parent Peer Support Providers' Self-Reported Fidelity to Peer Support | Baseline and 6 months later
  Parent peer support providers leading the virtual parent-led peer support groups will complete a self-reported measure related to rating their fidelity to peer support, outlining their adherence to peer support principles. The minimum score is 14, the maximum score is 70.

OTHER OUTCOMES:
Parent participant experiences | After 3 months in groups
  Virtual parent-led peer support group experiences of parents participants, qualitatively measured by semi-structured individual interviews with parents after 3 months in virtual parent-led peer support groups.
Parent Peer Support Provider experiences | After 6 months leading groups
  Virtual parent-led peer support group experiences of parent peer support providers, qualitatively measured by semi-structured focus group with virtual parent-led peer support groups and a focus group with parent peer support providers after 6 months of leading groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Couturier, MD MSc, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No